CLINICAL TRIAL: NCT01262729
Title: Xenon and Therapeutical Hypothermia After Successful Cardiopulmonary Resuscitation
Acronym: 10-015
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Feasibility and Recruitment problems
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Xenon-MTH-Study; 2010-022679-71 (EudraCT Number)
Record Dates: First submitted 2010-12-16; First posted 2010-12-17 (Estimated); Last update posted 2015-09-23 (Estimated); Status verified 2015-09

CONDITIONS: Efficacy and Safety of Xenon Inhalation; Successful Cardiopulmonary Resuscitation; Addition to Therapeutical Hypothermia
Keywords: xenon inhalation; therapeutical hypothermia; patients after cardiopulmonary resuscitation; efficacy; safety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Xenon-Arm (Experimental): Patients in Xenon-Arm will be inhalated with xenon within 2 hours additionally to therapeutical hypothermia after successful cardiopulmonary resuscitation.
  Interventions: Procedure: therapeutical hypothermia; Drug: Xenon Inhalation
- MTH (Active Comparator): Patients after successful cardiopulmonary resuscitation will be treated only with therapeutical hypothermia
  Interventions: Procedure: therapeutical hypothermia

INTERVENTIONS:
Procedure: therapeutical hypothermia — Patients after successful cardiopulmonary resuscitation will be treated in accordance to international guidelines (Guidelines 2005 on cardiopulmonary resuscitation. Resuscitation 2005; 67: S7-S23)
Drug: Xenon Inhalation — Patients after successful cardiopulmonary resuscitation will be inhalated with 65-70% Xenon within 2 hours additional to therapeutical hypothermia
  Arms: Xenon-Arm

SUMMARY:
In this clinical trial will be checked, whether 2 hour ventilation with xenon has neuroprotective effects in patients with out of hospital cardiac arrest and successful cardiopulmonary resuscitation

DETAILED DESCRIPTION:
Patients with out of hospital cardiac arrest and successful cardiopulmonary resuscitation will be randomized in two groups. First group (Treatment group) will be inhalated with xenon within 2 hours in addition to therapeutical hypothermia. The second group (Control group) will be treated with therapeutical hypothermia in accordance to international guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Patients with out of hospital cardiac arrest and successful cardiopulmonary resuscitation, which will be treated at Department of Internal Medicine I, University Hospital Aachen

Exclusion Criteria:

* Patients younger than 18 years
* Xenon allergy
* Pregnancy
* High expired oxygen requirement (>70%) in order to maintain adequate arterial oxygen saturation (SpO2>94%) at the beginning of treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2011-09; Primary Completion 2014-11 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Significant difference between treatment group and control group | within 28 days after cardiac arrest

SECONDARY OUTCOMES:
Safety and efficacy of xenon ventilation within 2 hours after successful cardiopulmonary resuscitation | within 28 days after cardiac arrest

CONTACTS AND LOCATIONS:
Overall Officials: Michael Fries, PD Dr. med., Principal Investigator — Surgical Intensive Care - Adults, University Hospital Aachen
Locations (1):
- Surgical Intensive Care - Adults, University Hospital Aachen, Aachen, North Rhine-Westphalia, Germany

REFERENCES:
- [Derived] Fries M, Brucken A, Cizen A, Westerkamp M, Lower C, Deike-Glindemann J, Schnorrenberger NK, Rex S, Coburn M, Nolte KW, Weis J, Rossaint R, Derwall M. Combining xenon and mild therapeutic hypothermia preserves neurological function after prolonged cardiac arrest in pigs. Crit Care Med. 2012 Apr;40(4):1297-303. doi: 10.1097/CCM.0b013e31823c8ce7. PMID 22425822